CLINICAL TRIAL: NCT00005815
Title: A Phase I/II Study of Temozolamide and Thalidomide in the Treatment of Advanced Melanoma
Brief Title: Temozolomide and Thalidomide in Treating Patients With Stage III or Stage IV Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 99-103; CDR0000067818 (Registry Identifier: PDQ (Physician Data Query)); NCI-G00-1786
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Intraocular Melanoma; Melanoma (Skin)
Keywords: iris melanoma; ciliary body and choroid melanoma, small size; ciliary body and choroid melanoma, medium/large size; extraocular extension melanoma; recurrent intraocular melanoma; stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — Temozolomide; Thalidomide

INTERVENTIONS:
Drug: temozolomide
Drug: thalidomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Thalidomide may stop the growth of melanoma by stopping blood flow to the tumor. Combining chemotherapy with thalidomide may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness temozolomide plus thalidomide in treating patients who have stage III or stage IV melanoma that cannot be removed during surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose (MTD) of temozolomide using an extended continuous schedule in combination with thalidomide in patients with advanced melanoma.
* Determine the response rate to this combination using an extended continuous schedule at the MTD in 30 patients who have advanced metastatic melanoma without brain metastases and in 15 patients who have metastatic melanoma in the brain.
* Further characterize the safety and toxicity of this combination in these patients.

OUTLINE: This is a dose escalation study of temozolomide (phase I) followed by a response rate determination study (phase II).

Patients receive oral temozolomide daily for 6 weeks followed by 2-4 weeks of rest. Patients receive oral thalidomide daily for the entire 8-10 week course. Treatment continues in the absence of unacceptable toxicity or disease progression.

Cohorts of 3-6 patients receive escalating doses of temozolomide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicities. Once the MTD is determined, additional patients are accrued to receive treatment with temozolomide and thalidomide at the recommended phase II dose.

PROJECTED ACCRUAL: A total of 3-24 patients will be accrued for phase I and then an additional 45 patients (15 with CNS disease, 30 without CNS disease) will be accrued for phase II of this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic malignant melanoma that is considered unresectable

  * Stage III or IV ocular, mucosal, or cutaneous melanoma
* Measurable disease
* No CNS disease (phase I only)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 150,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT/SGPT no greater than 3 times ULN
* Alkaline phosphatase no greater than 3 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No history of active angina
* No myocardial infarction within past 6 months
* No history of significant ventricular arrhythmia requiring medication with antiarrhythmics

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 4 weeks before and after study
* No frequent vomiting or medical condition that could interfere with oral medication intake (e.g., partial bowel obstruction)
* No preexisting neurotoxicity grade 2 or greater
* No serious concurrent infections treated with antibiotics
* No nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this study
* No psychiatric disorders that would preclude study compliance
* No other medical condition or reason that would preclude study
* No other malignancy within the past 2 years except:

  * Nonmelanoma skin cancer
  * Carcinoma in situ of the cervix
  * History of T1a or b prostate cancer detected incidentally at TURP and comprising less than 5% of resected tissue with PSA normal since TURP
* No AIDS related illness
* HIV negative

PRIOR CONCURRENT THERAPY:

* Recovered from prior therapy

Biologic therapy:

* At least 4 weeks since prior biologic therapy
* At least 4 weeks since prior immunotherapy
* No concurrent immunotherapy

Chemotherapy:

* No prior systemic chemotherapy for metastatic melanoma
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy, interstitial brachytherapy, or radiosurgery
* At least 3 weeks since prior radiotherapy to the brain if brain metastases from melanoma
* Prior radiotherapy to only indicator lesion allowed provided recent evidence of disease progression at that site
* No concurrent radiotherapy

Surgery:

* At least 2 weeks since prior surgery requiring general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-12; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Jen Hwu, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Hwu WJ, Krown SE, Menell JH, Panageas KS, Merrell J, Lamb LA, Williams LJ, Quinn CJ, Foster T, Chapman PB, Livingston PO, Wolchok JD, Houghton AN. Phase II study of temozolomide plus thalidomide for the treatment of metastatic melanoma. J Clin Oncol. 2003 Sep 1;21(17):3351-6. doi: 10.1200/JCO.2003.02.061. PMID 12947072
- [Result] Hwu WJ, Krown SE, Panageas KS, Menell JH, Chapman PB, Livingston PO, Williams LJ, Quinn CJ, Houghton AN. Temozolomide plus thalidomide in patients with advanced melanoma: results of a dose-finding trial. J Clin Oncol. 2002 Jun 1;20(11):2610-5. doi: 10.1200/JCO.2002.09.034. PMID 12039921